CLINICAL TRIAL: NCT01426269
Title: Evaluation of Relapse, Efficacy and Safety of Long-term Treatment With Oracea® Capsules Compared to Placebo After an Initial 12 Week Treatment Regimen With Oracea® and MetroGel® 1% in Adults With Rosacea
Brief Title: Evaluation of Relapse, Efficacy and Safety of Long-term Treatment With Oracea® vs Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: US10183
Record Dates: First submitted 2011-08-26; First posted 2011-08-31 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2014-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will receive placebo during phase 2 (week 12 - week 52)
  Interventions: Drug: Placebo
- Doxycycline and Metronidazole (Other): Subjects will receive Oracea® (oral doxycycline 40 mg USP (30 mg immediate release and 10 mg delayed release beads)) and MetroGel® 1% (topical metronidazole) during phase 1 (baseline to week 12)
  Interventions: Drug: Doxycycline; Drug: Metronidazole
- Doxycycline (Active Comparator): Subjects will receive Oracea® (oral doxycycline 40 mg USP (30 mg immediate release and 10 mg delayed release beads)) during phase 2 (week 12 - week 52)
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — During phase 1 (baseline - week 12): Oracea (doxycycline 40 mg USP (30 mg immediate release & 10 mg delayed release beads)), oral, one capsule daily in the morning During phase 1 (baseline - week 12) and phase 2 (week 12 - week 52): Oracea (doxycycline 40 mg USP (30 mg immediate release & 10 mg delayed release beads), oral, one capsule daily in the morning
  Other Names: Oracea® Capsules 40 mg
  Arms: Doxycycline; Doxycycline and Metronidazole
Drug: Metronidazole — During Phase 1: MetroGel 1% (metronidazole 1% gel), topical, apply a thin layer once daily to the affected area
  Other Names: Metrogel 1%
  Arms: Doxycycline and Metronidazole
Drug: Placebo — During phase 2 (week 12 - week 52): placebo, oral, one capsule daily in the morning
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess relapse, efficacy and safety in subjects with rosacea during long-term treatment with either Oracea® or placebo, after an initial 12-week regimen of Oracea® and MetroGel® 1%.

DETAILED DESCRIPTION:
Adult subjects with moderate to severe papulopustular rosacea will receive Oracea® and MetroGel® 1% once daily during phase 1 (baseline to week 12) of the study. Subjects will be eligible to enter phase 2 of the study based upon improvements in the Investigator's Global Assessment (IGA) score. During phase 2, subjects will receive either Oracea® or placebo once daily for up to an additional 40 weeks. Subjects who relapse during phase 2 will be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged 18 to 80 years inclusive.
* Subject with papulopustular rosacea (11 to 40 papules or pustules) and an IGA of moderate or severe.
* For subjects using medications to treat a concurrent medical condition, type and dose must have been stable for at least 90 days prior to study entry.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning a pregnancy during the study.
* Subject has any other active dermatological condition on the face that may interfere with the conduct of the study.
* Subject uses or has recently used any medication which may interfere with the absorption, distribution, or elimination of study medications, or may interfere with the assessments of efficacy or safety of the study medications.
* Subject has a known allergy to any of the components of the study products, and/or a known hypersensitivity to tetracyclines or metronidazole.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (11):
- United States (11):
  - ATS Clinical Research, Santa Monica, California
  - Dadeland Dermatology, Coral Gables, Florida
  - Melissa L. F. Knuckles M.D., P.S.C., Corbin, Kentucky
  - Dermatology Specialists Research, Louisville, Kentucky
  - Melissa L. F. Knuckles M.D., P.S.C., Richmond, Kentucky
  - The Maryland Laser, Skin, and Vein Institute, LLC, Hunt Valley, Maryland
  - Grekin Skin Institute, Warren, Michigan
  - Hilary Baldwin, Brooklyn, New York
  - The Center for Dermatology at Linden Oaks, Rochester, New York
  - Brodell Medical, Inc., Warren, Ohio
  - Center for Dermatology and Laser Surgery, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were treated with doxycycline or placebo for 52 weeks (Period 2) after a 12 week treatment regimen of doxycycline and metronidazole (Period 1). Subjects who completed period 1 with clear/near clear IGA, or achieved at least a 2 grade IGA improvement were eligible for period 2 of the study.
Groups:
- Doxycycline and Metronidazole Regimen: Subjects will receive Oracea® (oral doxycycline 40 mg USP (30 mg immediate release and 10 mg delayed release beads)) and MetroGel® 1% (topical metronidazole) during phase 1 (baseline to week 12)
  Oral Doxycycline and Topical Metronidazole: During phase 1 (baseline - week 12): Oracea (doxycycline 40 mg USP (30 mg immediate release & 10 mg delayed release beads)), oral, one capsule daily in the morning and MetroGel 1% (metronidazole 1% gel), topical, apply a thin layer once daily to the affected area.
  After Period 1, subjects who meet criteria for phase 2 will be randomized to receive doxycycline or placebo during phase 2
- Oral Doxycycline: Subjects will receive Oracea® (oral doxycycline 40 mg USP (30 mg immediate release and 10 mg delayed release beads)) during phase 2 (week 12 - week 52)
  Oral Doxycycline: During phase 2 week 12 - week 52: Oracea (doxycycline 40 mg USP (30 mg immediate release & 10 mg delayed release beads)), oral, one capsule daily in the morning
Period: Period 1: 12 Weeks
Arm/Group | Doxycycline and Metronidazole Regimen | Oral Doxycycline | Placebo
Started | 235 | 0 | 0
Completed | 180 | 0 | 0
Not Completed | 55 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Withdrawal by Subject | 22 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Lost to Follow-up | 22 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Period: Eligibility for Period 2, Randomization
Arm/Group | Doxycycline and Metronidazole Regimen | Oral Doxycycline | Placebo
Started | 180 | 0 | 0
Completed | 130 | 0 | 0
Not Completed | 50 | 0 | 0
Not completed — Did not qualify | 42 | 0 | 0
Not completed — Qualified, opted out | 8 | 0 | 0
Period: Period 2: 40 Weeks
Arm/Group | Doxycycline and Metronidazole Regimen | Oral Doxycycline | Placebo
Started | 0 | 65 | 65
Completed | 0 | 27 | 18
Not Completed | 0 | 38 | 47
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 9 | 11
Not completed — Protocol Violation | 0 | 5 | 5
Not completed — Lost to Follow-up | 0 | 8 | 6
Not completed — Site closed | 0 | 6 | 5
Not completed — Relapsed | 0 | 9 | 18

BASELINE CHARACTERISTICS:
Population: The safety population included 235 enrolled subjects. However, Baseline demographics were based on the ITT population which included 230 subjects; 5 subjects were excluded from this population due to consent issues.
Groups:
- Period 1: Oral Doxycycline and Topical Metronidazole: Subjects will receive oral doxycycline and topical metronidazole during period 1 (12 weeks)
  Oral Doxycycline and Topical Metronidazole: period 1, Oracea (doxycycline 40 mg USP (30 mg immediate release & 10 mg delayed release beads)), oral, one capsule daily in the morning and MetroGel 1% (metronidazole 1% gel), topical, apply a thin layer once daily to the affected area
Arm/Group | Period 1: Oral Doxycycline and Topical Metronidazole
Number analyzed (Participants) | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 217
  More than one race | 5
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 186
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 230
Skin Type [Number; unit: participants]
  Dry | 40
  Normal | 50
  Oily | 38
  Combination | 102
FItzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type Classification Scale I, always burns easily; never tans II, always burns easily; tans minimally and with difficulty III, burns minimally; tans gradually and uniformly (light brown) IV, burns minimally; always tans well (moderate brown) V, rarely burns; tans very easily (dark brown) VI, never burns, tans very easily (black)
  participants
    I | 16
    II | 93
    III | 64
    IV | 42
    V | 15
    VI | 0
History of Rosacea [Mean (Standard Deviation); unit: years] | 4.4 (7.7)
Height [Mean (Standard Deviation); unit: inches] | 66.0 (3.8)
Weight [Mean (Standard Deviation); unit: pounds] | 180.2 (45.0)

OUTCOME MEASURES:

1. Primary Outcome: Period 2: Number of Subjects Who Relapsed
Description: Subjects who relapsed during phase 2 were discontinued. Relapse was defined as meeting any one of the following criteria:
  * A return to the baseline lesion count
  * A return to the baseline IGA score
  * The investigator determines that a change in rosacea treatment is warranted due to the subject's clinical condition. The numbers reported here are accumulative numbers for each arm.
Time Frame: Period 2 (40 weeks)
Measure: Number; unit: participants
Groups:
- Oral Doxycycline: Subjects will receive Oracea® (oral doxycycline 40 mg USP (30 mg immediate release and 10 mg delayed release beads)) during period 2 (40 weeks) after 12 weeks of treatment with oral docycycline and topical metronidazole.
  Oral Doxycycline: During period 2, Oracea (doxycycline 40 mg USP (30 mg immediate release & 10 mg delayed release beads)), oral, one capsule daily in the morning
- Placebo: Subjects will receive placebo during period 2 (40 weeks) after 12 weeks of treatment with oral docycycline and topical metronidazole.
  Placebo: During period 2, placebo, oral, one capsule daily in the morning
Arm/Group | Oral Doxycycline | Placebo
Number analyzed (Participants) | 65 | 65
participants
  Week 4 | 4 | 10
  Week 8 | 8 | 14
  Week 12 | 9 | 16
  Week 16 | 9 | 16
  Week 20 | 9 | 16
  Week 24 | 9 | 17
  Week 28 | 9 | 18
  Week 32 | 9 | 18
  Week 36 | 9 | 18
  Week 40 | 9 | 18

2. Secondary Outcome: Period 2: Investigator's Global Assessment Success
Description: The evaluator (investigator) assessed the severity of rosacea at baseline and each postbaseline visit using a 5 point Investigator's Global Assessment scale. Subjects scores were then dichotomized into success (clear or near clear score) or failure (mild, moderate, or severe score).
Time Frame: Period 2 (40 weeks)
Measure: Number; unit: participants
Arm/Group | Oral Doxycycline | Placebo
Number analyzed (Participants) | 65 | 65
participants
  Week 4 | 44 | 38
  Week 8 | 36 | 33
  Week 12 | 33 | 37
  Week 16 | 38 | 34
  Week 20 | 35 | 33
  Week 24 | 36 | 32
  Week 28 | 39 | 35
  Week 32 | 39 | 34
  Week 36 | 40 | 33
  Week 40 | 41 | 33

3. Secondary Outcome: Period 2: Clinician's Erythema Assessment
Description: The evaluator (investigator) assessed the severity of erythema at baseline and each postbaseline visit using a total erythema score. The erythema of 5 areas of the face (forehead, chin, nose, right cheek, left cheek) was scored using a 5 point Clinician's Erythema Assessment scale (0 = none, 1 = mild, 2 = moderate, 3 = significant, 4 = severe). The total of the 5 individual erythema scores scores was the total erythema score.
Time Frame: Period 2 (40 Weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Doxycycline | Placebo
Number analyzed (Participants) | 65 | 65
units on a scale
  Week 4 | 5.0 (3.1) | 5.6 (3.8)
  Week 8 | 4.9 (3.5) | 5.8 (3.9)
  Week 12 | 4.7 (3.4) | 5.3 (4.3)
  Week 16 | 4.7 (3.4) | 5.2 (3.8)
  Week 20 | 4.3 (3.4) | 5.5 (3.8)
  Week 24 | 4.4 (3.5) | 5.3 (3.8)
  Week 28 | 4.3 (3.5) | 5.3 (3.8)
  Week 32 | 4.2 (3.6) | 5.3 (3.9)
  Week 36 | 4.4 (3.6) | 5.3 (3.8)
  Week 40 | 4.4 (3.5) | 5.3 (3.9)

4. Secondary Outcome: Period 2: Inflammatory Lesion Count
Description: The evaluator (investigator or a designee) performed lesion counts at each postbaseline visit.
Time Frame: Period 2 (40 Weeks)
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Oral Doxycycline | Placebo
Number analyzed (Participants) | 65 | 65
lesions
  Week 4 | 2.8 (4.5) | 5.8 (8.7)
  Week 8 | 3.1 (4.1) | 4.3 (6.0)
  Week 12 | 3.0 (4.2) | 1.9 (2.7)
  Week 16 | 2.4 (4.0) | 2.3 (2.6)
  Week 20 | 2.1 (2.2) | 2.6 (3.1)
  Week 24 | 2.2 (2.7) | 2.9 (3.9)
  Week 28 | 2.2 (2.8) | 2.9 (4.0)
  Week 32 | 2.2 (3.0) | 2.4 (3.3)
  Week 36 | 2.5 (3.1) | 2.2 (3.0)
  Week 40 | 2.1 (2.6) | 1.6 (1.9)

5. Other Pre Specified Outcome: Period 1: Tolerability (Scaling)
Description: Scaling, dryness, and stinging/burning were graded at baseline and weeks 4, 8, and 12 for subjects taking oral doxycycline and topical metronidazole.
Time Frame: Period 1 (12 Weeks)
Measure: Number; unit: participants
Groups:
- Baseline; Week 4; Week 8; Week 12: Subjects will receive Oracea® (oral doxycycline 40 mg USP (30 mg immediate release and 10 mg delayed release beads)) and MetroGel® 1% (topical metronidazole) during phase 1 (baseline to week 12)
Arm/Group | Baseline | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 235 | 235 | 235 | 235
participants
  None | 103 | 136 | 139 | 143
  Mild | 85 | 58 | 44 | 23
  Moderate | 44 | 24 | 11 | 2
  Severe | 3 | 0 | 0 | 0
  Missing | 0 | 17 | 41 | 67

6. Other Pre Specified Outcome: Period 1: Tolerability (Stinging/Burning)
Description: as for outcome 5
Time Frame: Period 1 (12 Weeks)
Measure: Number; unit: participants
Arm/Group | Baseline | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 235 | 235 | 235 | 235
participants
  None | 90 | 135 | 139 | 143
  Mild | 71 | 51 | 44 | 19
  Moderate | 60 | 31 | 11 | 6
  Severe | 14 | 1 | 0 | 0
  Missing | 0 | 17 | 41 | 67

7. Other Pre Specified Outcome: Period 1: Tolerability (Dryness)
Description: as for outcome 5
Time Frame: Period 1 (12 Weeks)
Measure: Number; unit: participants
Arm/Group | Baseline | Week 4 | Week 8 | Week 12
Number analyzed (Participants) | 235 | 235 | 235 | 235
participants
  None | 76 | 106 | 120 | 125
  Mild | 89 | 78 | 61 | 37
  Moderate | 60 | 32 | 13 | 6
  Severe | 10 | 2 | 0 | 0
  Missing | 0 | 17 | 41 | 67

ADVERSE EVENTS:
Time Frame: Period 1 (12 weeks of treatment with oral doxycycline and topical metronidazole) and Period 2 (40 weeks of treatment with oral doxycycline or placebo)
Groups:
- Period 2: Oral Doxycycline: Subjects will receive oral doxycycline during period 2 (40 weeks) after 12 weeks of treatment with oral docycycline and topical metronidazole.
  Oral Doxycycline: period 2, Oracea (doxycycline 40 mg USP (30 mg immediate release & 10 mg delayed release beads)), oral, one capsule daily in the morning
- Period 2: Placebo: Subjects will receive placebo during period 2 (40 weeks) after 12 weeks of treatment with oral docycycline and topical metronidazole.
  Placebo: period 2, placebo, oral, one capsule daily in the morning
Arm/Group | Period 1: Oral Doxycycline and Topical Metronidazole | Period 2: Oral Doxycycline | Period 2: Placebo
Serious Adverse Events (participants affected / at risk) | 4/235 | 2/65 | 2/65
Other Adverse Events (participants affected / at risk) | 9/235 | 6/65 | 7/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Oral Doxycycline and Topical Metronidazole (N=235) | Period 2: Oral Doxycycline (N=65) | Period 2: Placebo (N=65)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Oral Doxycycline and Topical Metronidazole (N=235) | Period 2: Oral Doxycycline (N=65) | Period 2: Placebo (N=65)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Upper respiratory (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less